CLINICAL TRIAL: NCT00123357
Title: Measuring Health Related Quality of Life in Veterans With Stroke
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: STI 20-029
Record Dates: First submitted 2005-07-18; First posted 2005-07-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-01

CONDITIONS: Stroke; Quality of Life; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Approximately 11,000 veterans annually are hospitalized with a newly acquired incident stroke. Based on American Heart Association ratios of stroke incidence and prevalence, up to 80,000 veterans may be stroke survivors. The assessment of outcomes in stroke survivors is important for clinical practice and research, yet there is no consensus on the best measures of stroke outcome in either clinical practice or research. We have developed a new stroke-specific outcome measure, the Stroke Impact Scale (SIS), to capture physical function and other dimensions of health-related quality of life.

DETAILED DESCRIPTION:
Background:

Approximately 11,000 veterans annually are hospitalized with a newly acquired incident stroke. Based on American Heart Association ratios of stroke incidence and prevalence, up to 80,000 veterans may be stroke survivors. The assessment of outcomes in stroke survivors is important for clinical practice and research, yet there is no consensus on the best measures of stroke outcome in either clinical practice or research. We have developed a new stroke-specific outcome measure, the Stroke Impact Scale (SIS), to capture physical function and other dimensions of health-related quality of life.

Objectives:

The major research questions in this investigation are: 1) Does the SIS have concurrent and discriminate validity in a veteran stroke population when compared to the FIM, Rankin, and the SF-36V? 2) What effect does mode of administration have on response rates, bias, data quality, reliability and validity, SIS domain scores, and cost of data collection? 3) What factors differentiate responders and non-responders? 4) Will the SIS scores predict health care costs and utilization?

Methods:

Using ICD-9 discharge codes and electronic medical records, patients were screened for a valid diagnosis of stroke. At three months post-stroke, patients were randomly assigned to receive a mailed SIS instrument or SIS via telephone interview. At four months post-stroke, all respondents were evaluated using the Functional Independence Measure and SF-36V by telephone.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

No exclusion criteria.

Exclusion Criteria:

No exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean M. Reker, PhD RN BS, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO; Pamela W. Duncan, PhD MA BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- Kansas City VA Medical Center, Kansas City, MO, Kansas, Illinois, United States

REFERENCES:
- [Result] Hayes J, Vogel B, Reker DM. Factors associated with VHA costs of care for first 12 months after first stroke. J Rehabil Res Dev. 2008;45(9):1375-84. PMID 19319761
- [Result] Kwon S, Hartzema AG, Duncan PW, Min-Lai S. Disability measures in stroke: relationship among the Barthel Index, the Functional Independence Measure, and the Modified Rankin Scale. Stroke. 2004 Apr;35(4):918-23. doi: 10.1161/01.STR.0000119385.56094.32. Epub 2004 Feb 19. PMID 14976324
- [Result] Jia H, Uphold CR, Wu S, Reid K, Findley K, Duncan PW. Health-related quality of life among men with HIV infection: effects of social support, coping, and depression. AIDS Patient Care STDS. 2004 Oct;18(10):594-603. doi: 10.1089/apc.2004.18.594. PMID 15630787
- [Result] Duncan P, Reker D, Kwon S, Lai SM, Studenski S, Perera S, Alfrey C, Marquez J. Measuring stroke impact with the stroke impact scale: telephone versus mail administration in veterans with stroke. Med Care. 2005 May;43(5):507-15. doi: 10.1097/01.mlr.0000160421.42858.de. PMID 15838417
- [Result] Duncan PW, Reker DM, Horner RD, Samsa GP, Hoenig H, LaClair BJ, Dudley TK. Performance of a mail-administered version of a stroke-specific outcome measure, the Stroke Impact Scale. Clin Rehabil. 2002 Aug;16(5):493-505. doi: 10.1191/0269215502cr510oa. PMID 12194620
- [Result] Kwon S, Duncan P, Studenski S, Perera S, Lai SM, Reker D. Measuring stroke impact with SIS: construct validity of SIS telephone administration. Qual Life Res. 2006 Apr;15(3):367-76. doi: 10.1007/s11136-005-2292-2. PMID 16547774